CLINICAL TRIAL: NCT00704951
Title: P05532 Evaluation of Treatment and Prophylaxis of Invasive Fungal Infections (IFIs) in Immuncompromised Patients in Austria. Version 1, 08-Nov-2007.
Brief Title: Evaluation of Treatment and Prophylaxis of Invasive Fungal Infections in Immuncompromised Patients in Austria (Study P05532)(WITHDRAWN)
Status: Withdrawn | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: P05532
Record Dates: First submitted 2008-06-23; First posted 2008-06-25 (Estimated); Last update posted 2015-08-25 (Estimated); Status verified 2015-08

CONDITIONS: Mycoses
MeSH Terms: conditions — Mycoses | interventions — posaconazole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients: Immunosuppressed/Immunocompromised patients at high risk for invasive fungal infections
  Interventions: Drug: Posaconazole or alternative fungal treatment

INTERVENTIONS:
Drug: Posaconazole or alternative fungal treatment — Dosage of Posaconazole:
  Prophylactic dosing: 200mg tid (600mg/day) Treatment dosing: 400mg bid (800mg/day)

SUMMARY:
The purpose of this program is to determine the frequency of the use of Posaconazole in immunocompromised patients refractory to first line therapy receiving therapeutic treatment based on different pathogens in comparison to other antifungal therapy.

A further objective is to determine the frequency of the use of Posaconazole in immunocompromised patients receiving prophylactic treatment in comparison to other antifungal prophylaxis.

ELIGIBILITY:
Inclusion Criteria:

* Immunocompromised patients with refractory IFI
* Patients eligible for prophylactic treatment due to anticipated neutropenia for more than 7 days.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Immunosuppressed/Immunocompromised patients at high risk for invasive fungal infections
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-07; Primary Completion 2011-05 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Safety: adverse events | Depending on treatment modality every 2 to 4 weeks

SECONDARY OUTCOMES:
Baseline: Patient demographic data; Disease history; Underlying diseases; Diagnosis; Previous therapies; Environmental risk factors; Host factors Performance status | Depending on treatment modality every 2 to 4 weeks
Treatment and follow up period: Performance status; Medication; Duration of treatment; Frequency of infectious episodes; Management of infections | Depending on treatment modality every 2 to 4 weeks
Adverse events; Survival status | Depending on treatment modality every 2 to 4 weeks